CLINICAL TRIAL: NCT02578940
Title: A Phase 3, Open-label Study to Assess the Clinical Utility of Fluciclovine (18F) PET/CT in Patients With Prostate Cancer With Biochemical Recurrence After Radical Treatment
Brief Title: Fluciclovine (18F) PET/CT in biochemicAL reCurrence Of Prostate caNcer
Acronym: FALCON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Blue Earth Diagnostics (Industry)
Collaborators: Innovate UK (Other Government); Syne Qua Non Limited (Industry); IND 2 Results LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BED-004
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-09

CONDITIONS: Cancer of the Prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: PET Imaging study
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Single intravenous administration of 18F-Fluciclovine for PET Scan
  Interventions: Drug: 18F-Fluciclovine PET CT

INTERVENTIONS:
Drug: 18F-Fluciclovine PET CT — Radioligand for PET CT scanning
  Other Names: FACBC

SUMMARY:
The main aim is to assess the impact of using 18F-fluciclovine (as a PET imaging radiotracer) on the clinical and treatment decision required for managing patients with biochemically recurrent prostate cancer (BCR) who are being considered for salvage treatment with the intention of providing disease cure. Also, this study will consolidate the information regarding diagnostic performance of fluciclovine PET/CT in a large number of prospectively followed patients at several centres in the UK and assess the effect of PSA level on the likelihood of detecting cancer lesions by 18F-fluciclovine

DETAILED DESCRIPTION:
Proposed Research In the setting of growing single-centre evidence of superior diagnostic performance of 18F-fluciclovine PET/CT in BCR, our primary aim is to assess its clinical impact on treatment decisions in a multi-centre study in patients with BCR being considered for radical salvage treatment (with curative intent). In addition, we aim to further characterise its diagnostic performance, afforded by larger numbers of patients from multi-centre recruitment. We also aim to assess the effect of PSA level on probability of lesion detection by 18F-fluciclovine.

ELIGIBILITY:
Inclusion Criteria:

* The subject has had an original diagnosis of PCa and underwent radical curative therapy at least 3 months before enrolment, and has been diagnosed with biochemical recurrence (BCR) on the basis of:

  1. Post radical radiotherapy (RRT) / brachytherapy: Increase in PSA level ≥2.0 ng/mL above the nadir level after radiotherapy (RT) or brachytherapy (ASTRO-Phoenix criteria) [53], or
  2. Post radical prostatectomy (RP): EITHER two consecutive rises in PSA and final PSA >0.1ng/ml OR three consecutive rises in PSA., This definition is also applicable to subjects with PSA persistence post RP (where the PSA fails to fall to undetectable levels).

  i. In addition, the subject post RP, should have a PSA doubling time of ≤15 months OR PSA level ≥1.0 ng/mL at time of recruitment. The PSA doubling time will be calculated using the Memorial Sloan Kettering Cancer Center nomogram (http://www.mskcc.org/nomograms/prostate/psa-doubling-time), based on a minimum of two PSA levels within 12 months of screening, taken after the last recorded nadir PSA available at time of screening.
* The subject has not had previous recurrences of PCa, i.e. this is the first diagnosis of BCR.
* The subject is being considered for radical salvage therapy.
* The subject is able and willing to comply with study procedures, and signed, dated and timed informed consent is obtained before any study-related procedure is performed.
* The subject's Eastern Cooperative Oncology Group [ECOG] performance status 0-2.
* The subject should not have received androgen-deprivation therapy within 3 months of screening.
* The subject has a normal or clinically acceptable medical history and vital signs findings at screening (up to 14 days before administration of study drug).

Exclusion Criteria:

* The subject has been previously included in this study.
* The subject has received, or is scheduled to receive, another investigational medicinal product (IMP) from 1 month before to 1 week after administration of fluciclovine (18F) injection.
* The subject has known hypersensitivity to fluciclovine (18F) injection or any of its constituents.
* The subject has had a choline PET/CT scan within 3 months of the screening visit.
* The subject has bilateral hip prostheses.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2018-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fergus Gleeson, FRCP FRCR, Principal Investigator — The Oxford University Hospitals NHS Trust
Locations (7):
- United Kingdom (7):
  - Mount Vernon Cancer Centre, Mount Vernon Hospital, Northwood, Middlesex
  - Churchill Hospital, Oxford, Oxfordshire
  - Royal Marsden Hospital, Sutton, Surrey
  - St James Institute of Oncology, Leeds, Yorkshire
  - Greater Glasgow & Clyde NHS Trust, Glasgow
  - University College London Hospital, London
  - St Thomas' Hospital, London

REFERENCES:
- [Derived] Andriole GL, Scarsbrook AF, Savir-Baruch B; LOCATE/FALCON Study Groups. Impact of 18F-fluciclovine PET/CT on plans for androgen deprivation therapy in patients with biochemical recurrence of prostate cancer: data analysis from two prospective clinical trials. Urol Oncol. 2023 Jun;41(6):293.e1-293.e7. doi: 10.1016/j.urolonc.2023.04.004. Epub 2023 Apr 29. PMID 37121865
- [Derived] Scarsbrook AF, Bottomley D, Teoh EJ, Bradley KM, Payne H, Afaq A, Bomanji J, van As N, Chua S, Hoskin P, Chambers A, Cook GJ, Warbey VS, Han S, Leung HY, Chau A, Miller MP, Gleeson FV; FALCON study group. Effect of 18F-Fluciclovine Positron Emission Tomography on the Management of Patients With Recurrence of Prostate Cancer: Results From the FALCON Trial. Int J Radiat Oncol Biol Phys. 2020 Jun 1;107(2):316-324. doi: 10.1016/j.ijrobp.2020.01.050. Epub 2020 Feb 14. PMID 32068113
- [Derived] Cook GJR. Performance of 18F-fluciclovine PET/MR in the evaluation of osseous metastases from castration-resistant prostate cancer. Eur J Nucl Med Mol Imaging. 2020 Jan;47(1):16-17. doi: 10.1007/s00259-019-04540-z. Epub 2019 Oct 17. No abstract available. PMID 31624865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between 27 November 2015 (first patient, screening visit) and 22 June 2018 (last patient, completed) at seven sites (one did not enrol) in the UK.
Period: Overall Study
Arm/Group | Single Arm
Started | 109
Received 18F-fluciclovine | 104
Completed | 103
Not Completed | 6
Not completed — Screening failure | 5
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Arm/Group | Single Arm
Number analyzed (Participants) | 104
Age, Continuous [Median (Full Range); unit: years] | 67.0 [49 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 104
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 104
Height [Median (Full Range); unit: cm] | 176.0 [157 to 197]
Weight [Median (Full Range); unit: Kg] | 82.80 [56.0 to 134.0]
Body Mass Index [Median (Full Range); unit: kg/m^2] | 26.50 [19.6 to 42.3]

OUTCOME MEASURES:

1. Primary Outcome: Impact on Patient Treatment /Management
Description: The record of the revised management plan post fluciclovine (18F) PET/CT scan in comparison to the pre-scan intended management plan.
Time Frame: 1 month
Population: For the primary analysis population, of the 104 patients included in the EAS, 58 patients with a positive 18F fluciclovine scan and 46 patients with a negative 18F fluciclovine scan had a pre-18F fluciclovine PET/CT management plan.
Measure: Count of Participants; unit: Participants
Groups:
- 18F-Fluciclovine PET CT: Single intravenous administration of 18F-Fluciclovine for PET Scan
  18F-Fluciclovine PET CT: Radioligand for PET CT scanning
Arm/Group | 18F-Fluciclovine PET CT
Number analyzed (Participants) | 104
Participants
  Overall Evaluable Analysis Set: Patients with Revised Management Plan | 66
  Overall Evaluable Analysis Set: No Revision to Management Plan | 38
  Positive 18F-fluciclovine Scan: number analyzed (Participants) | 58
  Positive 18F-fluciclovine Scan: Patients with Revised Management Plan | 53
  Positive 18F-fluciclovine Scan: No Revision to Management Plan | 5
  Negative 18F-fluciclovine Scan: number analyzed (Participants) | 46
  Negative 18F-fluciclovine Scan: Patients with Revised Management Plan | 13
  Negative 18F-fluciclovine Scan: No Revision to Management Plan | 33

2. Secondary Outcome: Response Rate to Radical Salvage Therapy
Description: To establish the proportion of patients who have a sustained response to radical salvage therapy.
Time Frame: 7 months
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-fluciclovine PET CT
Number analyzed (Participants) | 104
Participants
  Salvage therapy all: number analyzed (Participants) | 56
  Salvage therapy all: Treatment response | 43
  Salvage therapy all: Stable disease | 5
  Salvage therapy all: Disease progression | 8
  Salvage therapy guided by 18F-fluciclovine: number analyzed (Participants) | 17
  Salvage therapy guided by 18F-fluciclovine: Treatment response | 15
  Salvage therapy guided by 18F-fluciclovine: Stable disease | 0
  Salvage therapy guided by 18F-fluciclovine: Disease progression | 2
  Salvage therapy not guided by 18F-fluciclovine: number analyzed (Participants) | 39
  Salvage therapy not guided by 18F-fluciclovine: Treatment response | 28
  Salvage therapy not guided by 18F-fluciclovine: Stable disease | 5
  Salvage therapy not guided by 18F-fluciclovine: Disease progression | 6

3. Secondary Outcome: PSA Threshold for Positive Lesion Detection by 18F Fluciclovine PET/CT in BCR
Description: PSA levels in relation to scan positivity were analysed to determine the optimal PSA threshold for detecting recurrent prostate cancer by 18F fluciclovine PET/CT
Time Frame: 1 month
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of Detection Rate
Arm/Group | 18F-Fluciclovine PET CT
Number analyzed (Participants) | 104
percentage of Detection Rate
  PSA Subgroup 0 to 0.2 (ng/mL): number analyzed (Participants) | 18
  PSA Subgroup 0 to 0.2 (ng/mL) | 33.3 [13.3 to 59.0]
  PSA Subgroup >0.2 to 0.5 (ng/mL): number analyzed (Participants) | 27
  PSA Subgroup >0.2 to 0.5 (ng/mL) | 25.9 [11.1 to 46.3]
  PSA Subgroup >0.5 to 1.0 (ng/mL): number analyzed (Participants) | 11
  PSA Subgroup >0.5 to 1.0 (ng/mL) | 36.4 [10.9 to 69.2]
  PSA Subgroup >1.0 to 2.0 (ng/mL): number analyzed (Participants) | 5
  PSA Subgroup >1.0 to 2.0 (ng/mL) | 20 [0.5 to 71.6]
  PSA Subgroup >2.0 to 5.0 (ng/mL): number analyzed (Participants) | 24
  PSA Subgroup >2.0 to 5.0 (ng/mL) | 91.7 [73.0 to 99.0]
  PSA Subgroup >5.0 to 10.0 (ng/mL): number analyzed (Participants) | 11
  PSA Subgroup >5.0 to 10.0 (ng/mL) | 90.9 [58.7 to 99.8]
  PSA Subgroup >10 (ng/mL): number analyzed (Participants) | 8
  PSA Subgroup >10 (ng/mL) | 100 [63.1 to 100.0]

4. Secondary Outcome: Safety of 18F Fluciclovine Injection in Patients Undergoing PET/CT.
Description: Safety was assessed from data on the occurrence of adverse events (AEs) and changes in clinical laboratory tests, vital signs, injection-site status and physical examination findings from the time of administration of 18F fluciclovine injection throughout the study period.
Time Frame: 1 month
Population: Treatment-emergent Adverse Events
Measure: Count of Participants; unit: Participants
Groups:
- Treatment-emergent Adverse Events: Number of Subject from SAS who experienced Treatment-emergent Adverse Events
Arm/Group | Treatment-emergent Adverse Events
Number analyzed (Participants) | 27
Participants
  TEAEs Unrelated | 18
  TEAEs Possibly | 8
  TEAEs Probably | 0
  TEAEs Definitely | 1

ADVERSE EVENTS:
Time Frame: As specified in the Statistical Analysis Plan, results are presented as only those treatment-emergent adverse events which occurred up to 42 days after the 18F fluciclovine administration
Arm/Group | 18F-Fluciclovine PET CT
All-Cause Mortality (participants affected / at risk) | 0/104
Serious Adverse Events (participants affected / at risk) | 1/104
Other Adverse Events (participants affected / at risk) | 31/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 18F-Fluciclovine PET CT (N=104)
Urinary tract obstruction (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18F-Fluciclovine PET CT (N=104)
APPLICATION SITE REACTION (General disorders) | 3 (3)
FATIGUE (General disorders) | 3 (3)
APPLICATION SITE ERYTHEMA (General disorders) | 1 (1)
CATHETER SITE BRUISE (General disorders) | 1 (1)
INJECTION SITE ERYTHEMA (General disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 4 (4)
DIZZINESS (Nervous system disorders) | 2 (2)
DYSGEUSIA (Nervous system disorders) | 2 (2)
HYPOAESTHESIA (Nervous system disorders) | 1 (1)
PAROSMIA (Nervous system disorders) | 1 (1)
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1 (1)
TREMOR (Nervous system disorders) | 1 (1)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 3 (3)
BIOPSY PROSTATE (Investigations) | 1 (1)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 (1)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
ORAL HERPES (Infections and infestations) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
POST PROCEDURAL CONTUSION (Injury, poisoning and procedural complications) | 1 (1)
MELANOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 (1)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1)
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)
NECK MASS (Musculoskeletal and connective tissue disorders) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT02578940/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT02578940/SAP_001.pdf